CLINICAL TRIAL: NCT04938908
Title: Efficacy and Safety of Systemic and Ophthalmic Probiotic on Microbiota, Immunological and Clinical Outcomes of Patients With Dry Eye Syndrome
Brief Title: Probiotic in Dry Eye Syndromes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mojtaba Heydari, Principal Investigator, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 97-01-104-18912
Record Dates: First submitted 2021-06-22; First posted 2021-06-25 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ophthalmic probiotic (Experimental): 1 active drop in each eye/ 5 hours plus oral placebo capsule, for 4 weeks
  Interventions: Drug: Ophthalmic Probiotic; Dietary Supplement: Oral Placebo Capsule
- Placebo (Placebo Comparator): 1 placebo drop in each eye/ 5 hours plus oral placebo capsule, for 4 weeks
  Interventions: Drug: Opthalmic Placebo; Dietary Supplement: Oral Placebo Capsule
- Opthalmic Probiotic + Oral Probiotic (Experimental): 1 active drop in each eye/ 5 hours plus oral probiotic capsule, for 4 weeks
  Interventions: Drug: Ophthalmic Probiotic; Dietary Supplement: Oral Probiotic Capsule
- Oral Probiotic (Experimental): 1 placebo drop in each eye/ 5 hours plus oral probiotic capsule, for 4 weeks
  Interventions: Drug: Opthalmic Placebo; Dietary Supplement: Oral Probiotic Capsule

INTERVENTIONS:
Drug: Ophthalmic Probiotic — Bacterial lysate of Lactobacillus sakei, hydroxypropylmethylcellulose (HPMC), boric acid, sodium chloride, purified water.
  Arms: Ophthalmic probiotic; Opthalmic Probiotic + Oral Probiotic
Drug: Opthalmic Placebo — Placebo contains complete formulation of the active drug except for bacterial lysate of Lactobacillus sakei (i.e. HPMC, boric acid, sodium chloride, purified water)
  Arms: Oral Probiotic; Placebo
Dietary Supplement: Oral Probiotic Capsule — Live Lactobacillus sakei (5 billion cfus) in hydroxypropylmethylcellulose hard capsule, with maltodextrin excipient
  Arms: Opthalmic Probiotic + Oral Probiotic; Oral Probiotic
Dietary Supplement: Oral Placebo Capsule — Hydroxypropylmethylcellulose hard capsule, filled with maltodextrin excipient
  Arms: Ophthalmic probiotic; Placebo

SUMMARY:
This study will evaluate efficacy and safety of systemic and ophthalmic probiotic from bacterial lysate of Lactobacillus sakei on microbiota, immunological and clinical outcomes of patients with Dry Eye Syndrome.

DETAILED DESCRIPTION:
The ocular surface is comprised of the cornea and its overlying tissue, the conjunctiva. The ocular surface is continuously exposed to the external environment and, therefore, to different microbial species. A resident ocular surface microbiota has been found in various studies. Although little is known so far, some elements of this microbiota and/or its metabolites could represent protective cofactosr in the pathogenesis of common ocular diseases.

On the other hand, the gut microbiota is known to influence host homeostasis in distal tissues, such as brain (gut-barin axis), lungs (gut-lungs axis) and skin (gut-skin axis). However, little is known about distal effects of the gut microbiota on the ocular surface.

In this study we sought to evaluate the efficacy and safety aspects of L.sakei as both ophtalmic probiotic lysate and oral live probiotic on Dry Eye Syndrome, using a factorial design, against placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* 18<age<60
* BCVA (Best Corrected Visual Acuity) >=9/10
* At least 2 subjective complaints compatible with dry eye
* TBUT (Tear Break-Up Time) <= 10 sec, Schirmer's test <= 10mm
* Signed informed consent, voluntary adherence to treatment

Exclusion Criteria:

* Pregnancy/breastfeeding
* Conjunctivitis
* Thyroid disease
* Diabetes
* Rheumatologic diseases including Sjogren's syndrome
* Neurologic conditions, including stroke, Bell's palsy, Parkinson's, trigeminal nerve problem
* Refractive surgery (LASIK or PRK)
* Other Eye Surgeries
* HSV Keratitis
* Medication/supplement use, including psychiatric medicines, OTC cold medicines, anti-histamines, beta-blockers, pain relievers, sleeping pills, diuretics, Hormones replacement, and oral contraceptives
* Chemical splashes / injuries to the eyes
* Contact lens use
* Environmental (dusty, windy, hot/dry)
* Any treatment for dry eye in previous 4 weeks (including lubricants, steroids, cyclosporine)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index | 4 weeks
  Subjective score

SECONDARY OUTCOMES:
Tear break up time (TBUT) | 4 weeks
  Slit exam
Schirmer test | 4 weeks
  physical exam using Schirmer strip
Ocular surface microbiota composition | 4 weeks
  measured by 16s rRNA method
Tear Interleukin level | 4 weeks
  measured by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center for Traditional Medicine and History of Medicine-Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heydari M, Kalani M, Ghasemi Y, Nejabat M. The Effect of Ophthalmic and Systemic Formulations of Latilactobacillus sakei on Clinical and Immunological Outcomes of Patients With Dry Eye Disease: A Factorial, Randomized, Placebo-controlled, and Triple-masking Clinical Trial. Probiotics Antimicrob Proteins. 2024 Jun;16(3):1026-1035. doi: 10.1007/s12602-023-10079-1. Epub 2023 May 31. PMID 37256485